CLINICAL TRIAL: NCT06001541
Title: A Web-based Program to Improve Chronic Illness Self-management by Engaging Patients and Informal Caregivers
Brief Title: Web-based Program to Improve Self-management Among Veterans-caregiver Dyads
Acronym: Web-SUCCEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-137
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Medical Conditions
Keywords: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized clinical trial to evaluate the effectiveness of web-SUCCEED (Web-based Self-management Using Collaborative Coping EnhancEment in Diseases), a theoretically-derived, dyadic, self-management program. Web-SUCCEED is designed to improve self-management by improving dyadic stress coping and strengthening collaboration and communication.21 Web-SUCCEED comprises: 1) a three-module, self-paced behavioral intervention that Veterans and caregivers complete individually (one audio/video module per week) on the web-SUCCEED website; 2) brief, staff-led telephone calls in which dyads participate simultaneously after each module; and 3) peer support via a study-specific discussion board. Dyads learn and practice cognitive behavioral skills to reduce individual and relationship stress; improve positive emotions; improve communication and collaboration; increase pleasant activities; and maintain behavior change.
Who Masked: Investigator
Masking Description: the PI will be blinded to randomization and outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-SUCCEED+Enhanced Usual Care (Experimental): web-SUCCEED, usual care, psychoeducational materials and resources for caregivers.
  Interventions: Behavioral: Web-SUCCEED
- Enhanced Usual Care (Active Comparator): Usual care, enhanced by psychoeducational materials and resources for caregivers.
  Interventions: Behavioral: Web-SUCCEED

INTERVENTIONS:
Behavioral: Web-SUCCEED — web-SUCCEED (Web-based Self-management Using Collaborative Coping EnhancEment in Diseases), a theoretically-derived, dyadic, self-management program.20,21 Web-SUCCEED is designed to improve self-management by improving dyadic stress coping and strengthening collaboration and communication.21 Web-SUCCEED comprises: 1) a three-module, self-paced behavioral intervention that Veterans and caregivers complete individually (one audio/video module per week) on the web-SUCCEED website; 2) brief, staff-led telephone calls in which dyads participate simultaneously after each module; and 3) peer support via a study-specific discussion board. Dyads learn and practice cognitive behavioral skills to reduce individual and relationship stress; improve positive emotions; improve communication and collaboration; increase pleasant activities; and maintain behavior change.

SUMMARY:
The majority of Veterans will suffer from at least one chronic illness, often at great emotional and personal cost. Self-management is critical to improving physical and emotional outcomes, and many chronically ill Veterans receive self-management assistance from an informal caregiver, and both Veterans and informal caregivers experience individual and interpersonal stress as they navigate this journey. Yet, current clinical practices are not designed to effectively support the needs of both Veterans and their informal caregiver. Furthermore, self-management practices often require in-person visits, limiting access for Veterans and informal caregivers who live in rural areas, those with a physical disability, or those with financial challenges. This project tests a web-based, self-guided, behavioral intervention that targets the stress coping needs of Veterans with chronic illness and their informal caregivers. Results from this study could provide an important solution to the problem of poor self-management, which complicates the lives and prognosis of many Veterans.

DETAILED DESCRIPTION:
Background: For the 80% of older Americans who have at least one chronic condition, sharing self-management responsibilities with caregivers (relatives or friends) predicts longevity, better health, better quality of life, and fewer hospitalizations. Caregivers often support patients in their self-management efforts. This can bring patients and caregivers closer but can also generate stress for both that can interfere with self-management. Yet, self-management programs rarely support the coping needs of patient-caregiver dyads.

Significance: There are more than 5 million caregivers of Veterans; 75% of older Veterans receive some caregiver support. Caregivers incur individual financial and emotional costs even as they provide unpaid care. Having an effective self-management strategy that addresses the needs of both can improve outcomes and quality of life for millions of Veterans who suffer from chronic illnesses and their caregivers. This project addresses the priorities "Long-term care and Caregiving," "Virtual Care/Telehealth," and "Access to Care" and is consistent with the legislative goals of the MISSION Act.

Innovation and Impact: This highly innovative proposal uses the novel concept that strengthening the interpersonal relationships between Veterans and caregivers can improve the self-management of chronic conditions. It challenges current clinical paradigms by addressing the collective stress coping needs of dyads. It is methodologically innovative because unlike many behavioral intervention trials, it assesses barriers and facilitators to plan for future implementation. The focus on technology-enabled tools is timely given how COVID19 has transformed care delivery. This project takes advantage of the unique capabilities of the VA health system to explore questions including robust caregiver support and virtual care programs.

Specific Aims: With investments from VA HSR&D, the investigators have developed and successfully pilot tested a new theoretically-derived technology called Web-based Self-care Using Collaborative Coping EnhancEment in Diseases (web-SUCCEED). We propose to conduct a randomized clinical trial comparing web-SUCCEED to an enhanced usual care (EUC) control. The investigators will conduct a formative evaluation guided by the Consolidated Framework of Implementation Research (CFIR) to accelerate future implementation.

1. Assess whether web-SUCCEED improves Veteran outcomes of self-management compared to EUC, 4 weeks and 6 months following randomization.

2a. Assess whether web-SUCCEED improves patient stress and quality of life. 2b. Assess whether web-SUCCEED improves caregiver stress, quality of life and caregiver burden.

2c. Examine communication, dyadic coping, mutuality, and relationship quality as mediators of primary and secondary outcomes (Aims 1, 2a, 2b).

3. Guided by CFIR, conduct a formative evaluation involving key stakeholder interviews to understand barriers and facilitators of future implementation.

Methodology: The investigators will recruit 280 cognitively intact Veterans from VA Palo Alto Health Care System who are managing at least one common chronic condition, and their caregivers. Veteran-caregiver dyads will be randomized 1:1 to web-SUCCEED or EUC. Veteran and caregiver assessments will take place at baseline, then again at 4 weeks and 6 months. The formative evaluation will be guided by CFIR and involve semi-structured interviews with clinical staff, providers, and facility leaders in Year 4.

Next Steps: The formative evaluation will set the investigators up for implementation studies to evaluate web-SUCCEED in a wider array of clinical settings and facilities. Existing operational partnerships will facilitate wider clinical implementation and moving research into practice. The innovative project, strong investigative team and operational partnerships will ensure a successful study that has the potential to shift clinical paradigms.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be medically eligible if they have been diagnosed with at least one common chronic condition considered responsive to outpatient management as defined by being on the AHRQ list of Patient Quality Indicators, which are conditions that are considered responsive to high quality outpatient care.
* The investigators will also include conditions that are disproportionately high among Veterans (pain, mental health conditions).
* Based on the pilot study, the investigators anticipate this to include:

  * musculoskeletal pain
  * cardiovascular disease
  * diabetes
  * kidney disease
  * depression
* Eligible participants will have at least one outpatient visit in the prior 12 months related to their diagnosis and have a primary caregiver who lives with the Veteran. Dyads will be excluded if either the Veterans or their caregiver:

  * 1) have an implantable cardioverter defibrillator
  * 2) are on hemodialysis
  * 3) have received an organ transplant or are waitlisted for one
  * 4) are undergoing chemotherapy or radiation for cancer
  * 5) have limited life expectancy as determined by the provider or hospice care
  * 6) have dementia or other major cognitive deficits
  * 7) have a substance use disorder (SUD), since supporting interpersonal relationships in SUDs require specialized training that is outside the scope of web-SUCCEED
  * 8) have a paid caregiver who provides 50% or more support to the Veteran
  * 9) are actively psychotic or suicidal. Due to content overlap, the investigators will exclude Veterans who have participated in the Stanford CDSMP program, and caregivers who have participated in the Building Better Caregiver program

Exclusion Criteria:

Dyads deemed eligible with these criteria will be further screened by the study staff for internet use, self-management distress, and interpersonal violence.

* a. Internet Use: The investigators will use the question that used in the pilot study, "How often do you use a computer?" The investigators will exclude dyads where either Veterans or caregivers answer "less than once a week."
* b. Self-management Distress: The investigators will screen Veterans and caregivers for self-management distress using the same two-item measure that have been used for the pilot study of web-SUCCEED:

  * 1) How overwhelmed do you feel by the demands of living with your [OR Veteran's] health condition(s)?
  * 2) How often do you feel that you are failing in your routine to manage your [OR Veteran's] health conditions?" Respondents rate items from 1 (Not a problem) to 6 (A very serious problem), and scores are added. Dyads will be eligible if both individuals score a minimum of 2 and at least one scores >3.
* c. Interpersonal Violence: Veterans and caregivers will be separately screened with the question, "How do you and [Veteran, caregiver] handle stressful conversations or conflict?" If needed, this will be followed up with: "In the last year, has it gotten physical or have there been threats of physical force?". If the answer to the last question is "yes", dyads will not be eligible. Dr. Trivedi will assess for immediate safety, provide local resources, and involve authorities if appropriate. In the investigators' experience, this is a low likelihood event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-care of Chronic Illness Inventory Change | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  The SC-CII is based on the Middle Range Theory of Self-care. [Across three 10-item scales, the SC-CII assesses self-care maintenance (i.e., health-promoting and illness-related behaviors such as treatment adherence), self-care monitoring (i.e., ability to track symptoms and signs of an illness such as shortness of breath), and self-care management (i.e., ability to take action to deal with symptoms such as taking a diuretic to relieve fluid build-up). Coefficient alphas of the 3 subscales are: self-care monitoring (.81), self-care management (.71), and self-care maintenance (.67) in testing with patients with common chronic conditions. Each scale is standardized to a score of 100, and scores of 70 or more on each scale indicate adequate self-management.

SECONDARY OUTCOMES:
PROMIS Profile-29 v2.0 | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  Common Data Element indexed in the PhenX Toolkit that measures quality of life.
Caregiver Reaction Assessment | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  Positive and negative caregiver experience.
Perceived Stress Scale | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  Self-reported stress measure from PROMIS, 10 items.

OTHER OUTCOMES:
Couples Illness Communication Scale | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  Self-reported measure of communication, 4 items.
Pittsburgh Sleep Quality Index | Baseline (pre intervention), 6 week (post intervention), 6 month (follow-up)
  Measure of self-reported sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ranak B Trivedi, PhD MA MS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No